CLINICAL TRIAL: NCT01373138
Title: Randomized, Open-Label, 2-Way Crossover, Bioequivalence Study of Desloratadine and Pseudoephedrine 5 mg/240 mg Extended-Release Tablet and Clarinex-D® 24-Hour (Reference) Following a 5 mg/240 mg Dose in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Desloratadine and Pseudoephedrine Sulfate Extended-release Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Vice President - Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 50630
Record Dates: First submitted 2011-06-10; First posted 2011-06-14 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2006-06

CONDITIONS: Healthy
Keywords: Bioequivalence; Desloratadine and pseudoephedrine; crossover
MeSH Terms: interventions — desloratadine; Pseudoephedrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desloratadine and pseudoephedrine ER tablets 5/240 mg (Experimental): Desloratadine and pseudoephedrine ER tablets 5/240 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Desloratadine and pseudoephedrine
- Clarinex D 24-hour (Active Comparator): Clarinex D-24 of Schering Corporation Inc USA
  Interventions: Drug: Desloratadine and pseudoephedrine

INTERVENTIONS:
Drug: Desloratadine and pseudoephedrine — Desloratadine and pseudoephedrine 5/240 mg
  Other Names: Clarinex D-24

SUMMARY:
This is an open label randomised, 2-way crossover, comparative bioequivalence study.

DETAILED DESCRIPTION:
The objective of this study was to compare the rate and extent of absorption of Dr. Reddy's Laboratories Ltd., India, desloratadine-pseudoephedrine and Schering Corporation, U.S.A.(Clarinex-D® 24-HOUR), desloratadine-pseudoephedrine, administered as a 1 x 5 mg/240 mg extended-release tablet under fasting conditions. The treatment phases were separated by a washout period of 14 days. 34 subjects(19 males and 15 females) were dosed and were enrolled in the study; 31 of these enrolled subjects completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, non-smoker, ≥18 and ≤45 years of age.
* Capable of consent.
* Medically healthy with clinically normal laboratory profile, vital signs and ECG.
* BMI ≥19.0 and ≤30.0.

Exclusion Criteria:

* Clinically significant illness or surgery within 4 weeks prior to dosing.
* Any clinically significant abnormality or abnormal laboratory test results found during medical screening.
* Any reason which, in the opinion of the Medical Sub-Investigator, would prevent the subject from participating in the study.
* Positive test for hepatitis B, hepatitis C, or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
* History of significant alcohol abuse or drug abuse within one year prior to the screening visit.
* Regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [1 Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
* Use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to the screening visit or positive urine drug screen at screening.
* History of allergic reactions to desloratadine, pseudoephedrine or other related drugs.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; examples of inhibitors: antidepressants (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to administration of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to dosing.
* Clinically significant history or presence of any gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g.diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Any clinically significant history or presence of neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric, or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption and hormonal contraceptives.
* Difficulty to swallow study medication.
* Use of any tobacco products in the 3 months preceding drug administration.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the Medical Sub-Investigator, could contraindicate the subject's participation in this study.

  ● A depot injection or an implant of any drug (other than hormonal contraceptives) within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows:
* 50 mL to 499 mL of whole blood within 30 days,
* more than 499 mL of whole blood within 56 days prior to drug administration.
* Hemoglobin lower than 140g/L for males and 125 g/L for females.
* History or known presence of narrow-angle glaucoma, urinary retention, renal impairment, coronary artery or ischemic heart disease, diabetes mellitus, prostatic hypertrophy and hyperthyroidism.
* Positive urine pregnancy test at screening.
* Breast-feeding subject.
* Female subjects of childbearing potential having unprotected sexual intercourse with any non-sterile male partner (i.e. male who has not been sterilized by vasectomy for at least 6 months) within 14 days prior to study drug administration. Acceptable methods of contraception are:
* intra-uterine contraceptive device (placed at least 4 weeks prior to study drug administration;
* condom or diaphragm + spermicide;
* hormonal contraceptives (starting at least 4 weeks prior to study drug administration).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2006-04; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Denis Audet, MD, Principal Investigator — SFBC Anapharm
Locations (1):
- SFBC Anapharm, Sainte-Foy (Quebec), Canada